CLINICAL TRIAL: NCT02240719
Title: Phase I Study of Everolimus + Bendamustine in Patients With Relapsed/Refractory Hematological Malignancies
Brief Title: Everolimus and Bendamustine Hydrochloride in Treating Patients With Relapsed or Refractory Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 637004; 637004 (Registry Identifier: UC Davis); CRAD001NUS235T; UCDCC#245 (Other: University of California, Davis); NCI-2014-01934 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — Everolimus; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus + Bendamustine (Experimental): Patients receive bendamustine hydrochloride IV over 30 minutes on days 1 and 2 and everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: bendamustine hydrochloride

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda

SUMMARY:
This phase I trial studies the side effects and the best dose of everolimus when given together with bendamustine hydrochloride in treating patients with cancer of the blood (hematologic cancer) that has returned after a period of improvement (relapsed) or did not get better with a particular treatment (refractory). Everolimus may prevent cancer cells from growing by blocking a protein that is needed for cell growth. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving everolimus together with bendamustine hydrochloride may be a better treatment for hematologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of everolimus when administered in combination with bendamustine (bendamustine hydrochloride) in defined hematologic malignancies.

II. To determine the safety and tolerability of administering everolimus in combination with bendamustine chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the efficacy of everolimus when administered in combination with bendamustine in adult patients with relapsed/refractory hematological malignancies.

OUTLINE: This is a dose-escalation study of everolimus.

Patients receive bendamustine hydrochloride intravenously (IV) over 30 minutes on days 1 and 2 and everolimus orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease
* Baseline hemoglobin level of > 7.0 g/dl
* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* All the patients need to have biopsy proven active disease at the time of clinical trial
* Eastern Cooperative Oncology Group performance status of =< 2 study entry
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 50,000/mm^3
* Calculated creatinine clearance > 40 ml/min or 24 hour urine
* Total bilirubin =< 2 x upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal
* International normalized ratio < 2

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Any severe and/or uncontrolled medical conditions
* Uncontrolled diabetes mellitus
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks of the start of everolimus
* Known hypersensitivity to everolimus or bendamustine
* Known central nervous system (CNS) disease (NHL, diffuse large B cell lymphoma [DLBCL])
* Recent major surgery within 14 days prior to cycle 1, day 1
* Taking strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors
* Received live attenuated vaccines
* Known sero-positive for active or past viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are sero-positive because of hepatitis B virus vaccine are eligible
* History of another primary malignancy
* History of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Pregnant or nursing (lactating) women
* Women of childbearing potential
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
MTD of everolimus, defined as the dose that produces dose-limiting toxicity (DLT) in =< 1/6 patients, determined by incidence of DLT graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE version 4.0) and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.

SECONDARY OUTCOMES:
Incidence and severity of adverse events as defined by the NCI CTCAE version 4.03 | Up to 30 days post-treatment
Response rates (complete response, partial response, stable disease) | Up to 30 days post-treatment
  Response rate among patients with measurable disease will be summarized by exact binomial confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States